CLINICAL TRIAL: NCT00383747
Title: A Double Blind Placebo Controlled Trial of the Effects of Transdermal Nicotine on Cognitive Function in Non-Smokers With and Without Schizophrenia
Brief Title: The Effects of Nicotine on Cognition in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other); North Suffolk Mental Health Association (Other)
Responsible Party: Principal Investigator, A. Eden Evins, PI, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 04T574; CORRC 07-2004 (Other: North Suffolk Mental Health Association CORRC)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia
Keywords: cognition; nicotine; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine Patch (Active Comparator)
  Interventions: Drug: transdermal nicotine patch
- Placebo Nicotine Patch (Placebo Comparator)
  Interventions: Drug: Transdermal Nicotine Patch

INTERVENTIONS:
Drug: transdermal nicotine patch — 14mg transdermal nicotine application
  Other Names: Nicoderm CQ patch
  Arms: Nicotine Patch
Drug: Transdermal Nicotine Patch — 14mg transdermal nicotine application
  Arms: Placebo Nicotine Patch

SUMMARY:
Patients with schizophrenia have a variety cognitive deficits and nicotine has been shown to normalize some of these deficits. The purpose of this study is to investigate the effects of nicotine on cognition in schizophrenia.We will evaluate the effects of transdermal nicotine compared with placebo for attentional impairments in non-smokers with schizophrenia and controls.

DETAILED DESCRIPTION:
We propose to test the efficacy and safety of transdermal nicotine for attention and working memory in outpatients with stable symptoms of schizophrenia treated with high potency antipsychotic medications that do not smoke cigarettes or use nicotine-containing products. This is a randomized, double-blind, placebo-controlled pilot study to determine whether transdermal nicotine, initiated in a clinic setting and dosed for four hours is safe and effective for improving attention and spatial working memory deficits in patients with schizophrenia. This is an add-on study, subjects will continue with their usual medications and treatments throughout.

Subjects are 30- non-smoking outpatients with stable treated schizophrenia and 30 normal controls who do not have a major mental illness and who are matched for age sex and parental education. Subjects are randomized to one of 2 groups for order of receiving active and placebo patch, using a computer generated random number sequence. Randomization is concealed using opaque envelopes. Assessors and subjects are blind to group allocation.

The primary outcome measure is d' measure on the CPT-IP following a 4 hour administration of the transdermal nicotine patch. Secondary outcome measures are performance on tasks assessing attention, numeric and visuospatial working memory, psychomotor ability, executive functioning and motivation for reward following nicotine patch administration.

Specific Aims

1. To evaluate the effectiveness of transdermal nicotine compared with placebo for attentional impairment in patients with schizophrenia

   Hypothesis 1.1: Subjects will demonstrate greater signal detection as measured by the d' (hits vs. false alarms) on the Continuous Performance Test Identical Pairs Version (CPT-IP) following 4-hour nicotine administration when compared with placebo administration.

   Hypothesis 1.2: Subjects will demonstrate decreased false alarms on the CPT-IP following 4-hour nicotine administration when compared with placebo administration.

   Hypothesis 1.3: Subjects will demonstrate decreased reaction time on the CPT-IP following 4- hour nicotine administration when compared with placebo administration.
2. To evaluate the effect of transdermal nicotine in patients with schizophrenia compared with normal matched controls

Hypothesis 2.1: Schizophrenia subjects will demonstrate greater improvement in signal detection as measured by the d' (hits vs. false alarms) on the Continuous Performance test identical pairs version(CPT-IP) following 4-hour nicotine administration when compared with normal controls.

Hypothesis 2.2: Schizophrenia subjects will demonstrate greater reduction in false alarms on the CPT-IP following 4-hour nicotine administration when compared with normal controls.

Hypothesis 2.3: Schizophrenia subjects will demonstrate decreased reaction time on the CPT-IP following 4- hour nicotine administration when compared with normal controls. Performance Test Identical Pairs Version

ELIGIBILITY:
Inclusion Criteria:

Patients:

* DSM IV diagnosis of schizophrenia,
* age 18 - 60 inclusive,
* able to provide informed consent,
* treated with antipsychotic medications at a stable dose for at least 4 weeks,
* not treated with an investigational medication in the past 30 days,
* WRAT-3 IQ raw score greater than or equal to 35,
* non smokers for more than 3 months*,
* normal or corrected to normal vision.

Non Smoking defined by:

1. Self report of not smoking a single cigarette in the past 3 months.
2. Salivary Cotinine level < 30 ng/ml at screening and on the day of testing
3. Expired air CO < 9ppm on the day of the testing

Inclusion Criteria:

Control Group:

* Age 18 - 60 inclusive,
* able to provide informed consent,
* not treated with an investigational medication in the past 30 days,
* WRAT-3 IQ raw score greater than or equal to 35,
* non smokers for more than 3 months*,
* normal or corrected to normal vision,
* Non Smoking as defined above.

Exclusion Criteria:

Patients:

* Use of any nicotine containing product in the past 3 months by self report,
* use of cholinesterase inhibitors such as galantamine in the past 3 months,
* untreated ischaemic heart disease,
* uncontrolled hypertension,
* current unstable serious medical illness (renal, neoplastic, hematological),
* allergy to patches.
* Currently or planning to be pregnant in the next 8 weeks, as verified by positive pregnancy test, or childbearing potential and not using adequate contraception. Those not of childbearing potential include post-menopausal, surgically sterilized, and male participants.
* Substance abuse in the past month: self-reported, diagnosed during chart review, and verified by a positive salivary test for cotinine, cocaine, methamphetamine, amphetamine, ethanol, TCH, opiates or PCP at screen.
* Recent deterioration in mental state, current major depressive disorder, history of cognitive impairment secondary to other disorders such as head injury, dementia, general medical condition, diagnosis of mental retardation

Exclusion criteria:

Controls:

* Past or present DSM IV diagnosis of schizophrenia, schizoaffective disorder, major depression, bipolar disorder, or mental retardation.
* First degree relative with diagnosis of schizophrenia or schizoaffective disorder,
* use of cholinesterase inhibitors such as galantamine in the past 3 months,
* untreated ischaemic heart disease,
* uncontrolled hypertension,
* current unstable serious medical illness (renal, neoplastic, hematological,)
* allergy to patches,
* currently or planning to be pregnant in the next 8 weeks, as verified by positive pregnancy test, or childbearing potential and not using adequate contraception. Those not of childbearing potential include post-menopausal, surgically sterilized, and male participants.
* Substance abuse in the past month: self-reported, diagnosed during chart review, and verified by a positive salivary test for cotinine, cocaine, methamphetamine, amphetamine, ethanol, TCH, opiates and PCP at screen.
* History of cognitive impairment secondary to other disorders such as head injury, dementia, general medical condition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2004-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A E EVINS, MD MPH, Principal Investigator — Massachusetts General Hosptal
Locations (1):
- Massachusetts General Hospital Schizophrenia Research Program, Boston, Massachusetts, United States

REFERENCES:
- [Result] Barr RS, Culhane MA, Jubelt LE, Mufti RS, Dyer MA, Weiss AP, Deckersbach T, Kelly JF, Freudenreich O, Goff DC, Evins AE. The effects of transdermal nicotine on cognition in nonsmokers with schizophrenia and nonpsychiatric controls. Neuropsychopharmacology. 2008 Feb;33(3):480-90. doi: 10.1038/sj.npp.1301423. Epub 2007 Apr 18. PMID 17443126
- [Result] Barr RS, Pizzagalli DA, Culhane MA, Goff DC, Evins AE. A single dose of nicotine enhances reward responsiveness in nonsmokers: implications for development of dependence. Biol Psychiatry. 2008 Jun 1;63(11):1061-5. doi: 10.1016/j.biopsych.2007.09.015. Epub 2007 Nov 5. PMID 17976537
- [Result] Jubelt LE, Barr RS, Goff DC, Logvinenko T, Weiss AP, Evins AE. Effects of transdermal nicotine on episodic memory in non-smokers with and without schizophrenia. Psychopharmacology (Berl). 2008 Jul;199(1):89-98. doi: 10.1007/s00213-008-1133-8. Epub 2008 Jun 12. PMID 18548234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-smoking adults with a DSM IV diagnosis of schizophrenia or schizoaffective disorder, depressed type, were recruited from an urban community mental health clinic. Non-smoking adults without psychiatric illness were recruited using advertising in local press and internet sites. All study procedures took place between January 2005 and July 2006.
Pre-assignment Details: Once enrolled, participants attended a baseline visit followed by 2 study days. At the first visit, subjects underwent a training session in the Cognitive Drug Research battery and subjects with schizophrenia completed baseline clinical scales including the Scale for Assessment of Negative Symptoms (SANS) and Positive and Negative Syndrome Scale
Groups:
- Non-smokers w/Schizophr: Nicotine Patch (V1) Then Placebo (V2): Nonsmokers with schizophrenia on a stable dose of antipsychotic medication received first transdermal nicotine patch: 14mg transdermal nicotine application then placebo patch
- Nonsmokers w/Schizophr: Placebo (V1) Then Nicotine Patch (V2): Non smokers with schizophrenia received Placebo patch application then Nicotine patch: 14mg transdermal nicotine
- Controls: Nicotine Patch (V1) Then Placebo (V2): Non-smoking adults without psychiatric illness received transdermal nicotine patch: 14mg transdermal nicotine application then placebo patch
- Controls: Placebo (V1) Then Nicotine Patch (V2): Non-smoking adults without psychiatric illness received placebo patch then nicotine patch 14mg transdermal nicotine application
Period: Visit 1
Arm/Group | Non-smokers w/Schizophr: Nicotine Patch (V1) Then Placebo (V2) | Nonsmokers w/Schizophr: Placebo (V1) Then Nicotine Patch (V2) | Controls: Nicotine Patch (V1) Then Placebo (V2) | Controls: Placebo (V1) Then Nicotine Patch (V2)
Started | 14 | 14 | 16 | 16
Completed | 14 | 14 | 16 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Visit 2
Arm/Group | Non-smokers w/Schizophr: Nicotine Patch (V1) Then Placebo (V2) | Nonsmokers w/Schizophr: Placebo (V1) Then Nicotine Patch (V2) | Controls: Nicotine Patch (V1) Then Placebo (V2) | Controls: Placebo (V1) Then Nicotine Patch (V2)
Started | 14 | 14 | 16 | 16
Completed | 14 | 14 | 16 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non Smokers With Schizophrenia | Controls | Total
Number analyzed (Participants) | 28 | 32 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (8) | 40 (11) | 43 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Effects of Nicotine Patch Compared With Placebo in Non- Smokers With Schizophrenia and Control Groups on Attention Measured by the Continuous Performance Test Identical Pairs Version
Description: The primary outcome measure was attention as measured by the Continuous Performance Test Identical Pairs (CPT-IP) Version 4.0 (Biobehavioral Technologies, New York, USA), developed for use in patients with schizophrenia and normal controls. In this task, participants were asked to respond when two identical pairs of numbers were presented in sequence by pressing a mouse key as quickly as possible using the dominant hand.The stimuli were presented with increasing cognitive load in successive blocks: two-,three- and four-digit target in the first, second and third block, respectively. Hit reaction time, a standard outcome variables on the CPTIP, is presented here. It was measured 3 hrs after application of the patch
Time Frame: Visit 1 and visit 2 (separated by an interval of 7-10 days)
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Non Smokers With Schizophrenia + Nicotine Patch: Nonsmokers with schizophrenia on a stable dose of antipsychotic medication + transdermal nicotine patch: 14mg transdermal nicotine application
- Non Smokers With Schizophrenia + Placebo Nicotine Patch: Non smokers with schizophrenia + Placebo transdermal nicotine patch: 14mg transdermal nicotine application
- Control + Nicotine Patch: Non-smoking adults without psychiatric illness + transdermal nicotine patch: 14mg transdermal nicotine application
- Controls + Placebo Nicotine Patch: Non-smoking adults without psychiatric illness + placebo transdermal nicotine patch: 14mg transdermal nicotine application
Arm/Group | Non Smokers With Schizophrenia + Nicotine Patch | Non Smokers With Schizophrenia + Placebo Nicotine Patch | Control + Nicotine Patch | Controls + Placebo Nicotine Patch
Number analyzed (Participants) | 28 | 28 | 32 | 32
milliseconds | 2.2 (0.8) | 2.1 (0.8) | 3.4 (0.6) | 3.2 (0.6)

2. Secondary Outcome: Effects of Nicotine Patch Compared With Placebo in Non- Smokers With Schizophrenia and Control Groups on Visual Attention and Cognitive Interference as Measured by Three Card Stroop
Description: This standard test of visual attention, processing speed and cognitive interference was performed, in which three cards (Stoelting Co., Wood Dale, IL, USA) were presented in order: the first card with color names, the second with colored patches of ink and the third with color namesprinted in incongruously colored ink. Participants were asked to read or name as many colors as possible in 45 s for each condition. The raw interference score was calculated by subtracting the predicted color-word score (calculated using raw word and color scores) from the observed raw color-word score. This value was converted to an interference T score by referring to a standardized table. A higher interference T score indicates better task performance with less interference. It was measured 3 hrs after application of the patch, after CPT
Time Frame: Visit 1 and visit 2 (separated by an interval of 7-10 days)
Measure: Mean (Standard Deviation); unit: score
Groups:
- Non-smokers With Schizophrenia + Nicotine Patch: Nonsmokers with schizophrenia on a stable dose of antipsychotic medication received first transdermal nicotine patch: 14mg transdermal nicotine application
- Nonsmokers With Schizophrenia +, Placebo: Non smokers with schizophrenia received Placebo patch application
- Control + Nicotine Patch: Non-smoking adults without psychiatric illness received transdermal nicotine patch: 14mg transdermal nicotine application
- Control + Placebo: Non-smoking adults without psychiatric illness received placebo patch
Arm/Group | Non-smokers With Schizophrenia + Nicotine Patch | Nonsmokers With Schizophrenia +, Placebo | Control + Nicotine Patch | Control + Placebo
Number analyzed (Participants) | 28 | 28 | 32 | 32
score | 50.4 (5.8) | 49.0 (4.6) | 56.8 (10.3) | 58.8 (10.0)

3. Secondary Outcome: Effects of Nicotine Patch Compared With Placebo in Non- Smokers With Schizophrenia and Control Groups on Letter Number Sequencing
Description: This measure of working memory and auditory attention was performed under two conditions. In the first condition, participants were read progressively longer lists of letters and numbers and instructed to repeat these exactly as given, without reordering. In the second condition, participants were read progressively longer lists of numbers and letters and instructed to re-order the list and give the numbers first in ascending order and then the letters in alphabetical order (WMS-III). The sum of the trial scores provided the item score and the sum of the item scores provided the total score.It was measured 3 hrs after application of the patch, after CPT and Stroop. The total score ranges from 0 to 21.Higher scores of Letter number sequencing means better working memory and auditory attention
Time Frame: Visit 1 and visit 2 (separated by an interval of 7-10 days)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nonsmokers With Schizophrenia + Placebo: Non smokers with schizophrenia received Placebo patch application
Arm/Group | Non-smokers With Schizophrenia + Nicotine Patch | Nonsmokers With Schizophrenia + Placebo | Control + Nicotine Patch | Control + Placebo
Number analyzed (Participants) | 28 | 28 | 32 | 32
units on a scale
  without reorder | 12.6 (3.3) | 12.5 (3.4) | 15.5 (3.3) | 15.9 (3.4)
  with reorder | 8.8 (3.1) | 9.0 (2.6) | 12.2 (3.4) | 12.6 (3.1)

4. Secondary Outcome: Effects of Nicotine Patch Compared With Placebo in Non- Smokers With Schizophrenia and Control Groups on Lateralized Psychomotor Speed Measured by the Grooved Pegboard
Description: The Grooved Pegboard (model 32025 Lafayette Instrument Company, Lafayette, IN, USA). In this test of lateralized psychomotor speed, participants had 45 s to place as many pegs as possible into grooves on a board using their dominant hand. The number of correctly placed pegs were recorded for each of the two trials.It was measured 3 hrs after application of the patch after CPT, Stroop and Letter number sequencing
Time Frame: Visit 1 and visit 2 (separated by an interval of 7-10 days)
Measure: Mean (Standard Deviation); unit: number of pegs into grooves
Arm/Group | Non-smokers With Schizophrenia + Nicotine Patch | Nonsmokers With Schizophrenia + Placebo | Control + Nicotine Patch | Control + Placebo
Number analyzed (Participants) | 28 | 28 | 32 | 32
number of pegs into grooves | 14.4 (3.6) | 14.5 (3.2) | 19.1 (3.2) | 18.6 (2.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at every visit
Arm/Group | Non Smokers With Schizophrenia | Controls
Serious Adverse Events (participants affected / at risk) | 2/28 | 0/32
Other Adverse Events (participants affected / at risk) | 3/28 | 6/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Smokers With Schizophrenia (N=28) | Controls (N=32)
allergic reaction to peanuts (Immune system disorders) | 1 (1) | 0 (0)
deterioration in mental state (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Non Smokers With Schizophrenia (N=28) | Controls (N=32)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4)
skin irritations (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) — Mild adverse events have been reported in aggregate, unblinded data is not available at this point. Mild adverse events included minor skin irritations (17 subjects)
Dizziness (Nervous system disorders) | 0/0 (0) | 0/0 (0) — Mild adverse events have been reported in aggregate, unblinded data is not available at this point. Mild adverse events also included dizziness (14 subjects)
Headache (General disorders) | 0/0 (0) | 0/0 (0) — Mild adverse events have been reported in aggregate, unblinded data is not available at this point. Mild adverse events also included headache (11 subjects)
Palpitations (General disorders) | 0/0 (0) | 0/0 (0) — Mild adverse events have been reported in aggregate, unblinded data is not available at this point. Mild adverse events also included palpitations (seven subjects).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No